CLINICAL TRIAL: NCT01000103
Title: Using Repetitive Transcranial Magnetic Stimulation (rTMS) in the Rehabilitation of Chronic Spatial Neglect After Stroke: A Double Blind Study
Brief Title: Using Repetitive Transcranial Magnetic Stimulation (rTMS) in the Rehabilitation of Chronic Spatial Neglect After Stroke
Acronym: NEGLECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P071238; ID RCB 2009-A00280-57 (Other: ID RCB 2009-A00280-57)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Cerebrovascular Disorders; Cerebral Stroke; VISIO-spatial Neglect; VISUO-spatial Extinction
Keywords: Stroke; Visuospatial neglect; Visuospatial extinction; Transcranial Magnetic Stimulation (TMS); Non-invasive brain stimulation; Neuromodulation; Brain parietal cortex; Neurological sequels; Cognitive rehabilitation
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Real rTMS treatment (Active Comparator): Transcranial Magnetic Stimulation, in a low frequency (1 Hz) continuous train of 20 minutes (1200 pulses)
  Interventions: Device: Real rTMS
- 2: Sham rTMS treatment (Sham Comparator): Simulation of rTMS
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Real rTMS — Transcranial Magnetic Stimulation, in a low frequency (1 Hz) continuous train of 20 minutes (1200 pulses)
  Arms: 1: Real rTMS treatment
Device: Sham rTMS — two TMS coils will be used: a passive one which is placed flat on top of the "actively" targeted region which remains unplugged and generates a continuous scalp tactile sensation, and an active one located at a prudential distance from the scalp, which will deliver active pulses and its accompanying sensations
  Arms: 2: Sham rTMS treatment

SUMMARY:
Visuospatial neglect is a common neurological symptom which appears following strokes on regions of the right hemisphere of the brain. It affects patient's self representation and awareness of the space, impairing functional rehabilitation and adaptation back to a normal life. The primary purpose of this protocol is to assess the impact of 10 daily sessions of a non-invasive brain stimulation technique, low frequency repetitive Transcranial Magnetic Stimulation (rTMS), applied on the intact hemisphere of the brain to treat post stroke visuospatial neglect at the chronic stage. The hypothesis is that a regime of real but not sham rTMS on the left posterior parietal cortex of the brain will long-lastingly ameliorate visuospatial neglect in stroke patients as revealed by clinical paper-and-pencil and computer-based tests assessing search, detection and discrimination of stimuli presented in different areas of the visual field.

DETAILED DESCRIPTION:
Scientific aims and goals:

The long-term goal aim of this application is to provide evidence of the role of a non-invasive neuromodulation technique such as rTMS in the treatment of chronic neurological sequels generated after strokes in human patients. Such interventions are based in an "at will" modulation the level of activity in intact regions, resulting in an enhancement of excitatory projections or the suppression of inhibitory influences driven through spared connectivity. They result in activity increases of the stroke surviving neurons, allowing the re-emergence of function after brain damage. Such principles can be applied to different sorts of neurological sequels for which the underlying connectivity and its post-stroke status is well known. In this specific project, we propose the use of low frequency rTMS on the intact left posterior parietal cortex (in the intraparietal sulcus, IPS) to improve the symptoms of visuospatial neglect derived form right stroke injuries including the posterior parietal cortex. Such project is based in the interhemispheric rivalry hypothesis, according to which, spatial neglect is in part caused by the over inhibition exerted from the intact left parietal cortex onto the injured left homologue regions, which are mediated by well-known overall inhibitory transcallosal projections between the left and the right hemispheres. According to this hypothesis and preliminary data, the reduction of the left parietal disinhibition should result into a lesser degree of suppression exerted by the intact left hemisphere sites onto the right injured parietal areas, process which will along the emergence of activity.In this context, we defined a primary aim accompanied by two secondary aims, which will be tackled in parallel:Primary AIMS AIM1: To assess the effects of repetitive Transcranial Magnetic Stimulation (rTMS) in the treatment of chronic visuospatial neglect generated by stroke Secondary AIMS AIM 2: To assess the durability of such a recovery over time once the treatment is completed and discontinued AIM 3: To further assess the safety of such therapeutic approach based in the deactivation of an intact -but hyperexcited region- holding connectivity with the damaged area.

Evaluation criteria Main criteria -Changes in the Spatial Bias Compound Score (SBCS) between pre (baseline) and post 10 days of rTMS treatment Such score is calculated on the basis of the result of 4 subtests which include: (1) bells cancellation task, (2) a copy of the GAINOTTI figure, (3) identification of overlapping figures, and (4) line bisection, according to the following formula (SBCS=λ=ln(XR/XL), considering the identification or copying of elements presented on the right or the left visual fields of the patient. The subtests of the SBCS will be also individually assessed and followed.

Secondary criteria

1. Efficacy criteria
2. Safety criteria
3. Predictive factors assessmentStudy population and duration of studyWe will study a population of stroke patients with chronic signs of hemispatial neglect with at least 3 months of evolution (n=148, 2 groups of 74 patients) recruited across 48 months at an approximate rate of 37 patients /year.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral right hemisphere stroke
2. Visuospatial neglect or extinction at the time of entry, as determined by at least 1 test of the battery (BEN) displaying pathological scores (cut off values as defined in AZOUVI et al. JNNP 2004, Table 1), or an ECB test, score > 8
3. A period of evolution of at least 3 months since stroke event
4. Age between 18 and 75 years old
5. Affiliation to Social Security system
6. Informed consent signature

Exclusion Criteria:

1. Criteria related to the stroke:

   * Bilateral stroke lesions: left hemispheric focal lesion excluding leucoaraiosis or mild lesions of the white matter
2. Criteria related to rTMS:

   * Metal in the head, or a history of prior neurosurgical procedures
   * Ferromagnetic bioimplants activated by any electronic, mechanical or magnetic means such as: cochlear implants, pacemakers, medication pumps, vagal stimulators, deep brain stimulators, neurostimulators, bio stimulators, or ventriculoperitoneal shunts.
   * Prior history of seizures or seizure events following the stroke requiring the use of antiepileptic drugs
   * Pregnancy (by history or positive urine pregnancy test)
   * A urine pregnancy test will be done on all women of childbearing potential (those who have started menstruating up until they have stopped menstruating) prior to each MRI session, to rule out pregnancy.
   * Diagnosis of tinnitus
   * Participation in any experimental neglect rehabilitation project for at least 5 weeks before and 2 weeks after the stimulation, or during the 6 months of follow-up.
   * Prior participation in TMS based treatments or experiments
3. Criteria related to feasibility:

   * Incapacity to follow and complete the stimulation and follow-up protocol
   * Other medical cerebral conditions other than the condition studied in the present protocol
   * Any general medical condition, which could potentially interfere with clinical progression
   * Any incapacitating psychiatric conditions, including significant history of substance abuse and severe depression
   * Chronic treatment with medications that might modify cortical excitability
   * Subjects with visual impediments that would limit our ability to obtain reliable testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-03-24 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

PRIMARY OUTCOMES:
Changes in the Spatial Bias Compound Score (SBCS). Such score is calculated on the basis of the result of 4 subtests | between pre (baseline) and post 10 days of rTMS treatment

SECONDARY OUTCOMES:
Changes in Catherine BERGEGO Scale and-or equivalent ecological test | between pre (baseline) and every subsequent evaluation
Changes in the percentage of correct target detections vs. total | between pre (baseline) and every subsequent evaluation
Changes in the Normalized reaction time of correct detections | between pre (baseline) and every subsequent evaluation
potential clinically relevant side-effect caused by the use of TMS in terms of neurological manifestations such as: seizure, occurrence of additional stroke, or signs of enhanced intracranial pressure. | During rTMS treatment and the 6 months follow-up
changes in cognitive functions processed by the intact left parietal cortex | between baseline and every subsequent evaluation, during the 6 months follow-up
Changes of the main cognitive domains and depression status according to the Mini-Mental test and Hamilton depression scale | between pre (baseline) and every subsequent evaluation
Correlation between treatment efficacy and lesion location and extent | Any time after the end of rTMS treatment
Correlation between treatment efficacy and severity of Neglect and other associated clinical deficits | Any time after the end of rTMS treatment
Correlation between treatment efficacy and rTMS parameters and patient's cortical excitability and sensations | Any time after the end of rTMS treatment
Correlation between treatment efficacy and daily activities with potential impact on Neglect | Any time after the end of rTMS treatment
Evaluation of SBCS and its subscores at each follow-up visits | 5 days, 10 days, 15 days, 20 days, 27 days, 40 days, 70 days, 130 days and 190 days after 1st rTMS session.
Changes in neurological conditions according to: Rankin, Barthel and NIH SS scores | Between baseline and every subsequent evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pascale PRADAT-DIEHL, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Antoni VALERO-CABRE, MD-PhD, Principal Investigator — Centre National de la Recherche Scientifique, France
Locations (1):
- Hôpital de la Salpétrière, Paris, France